CLINICAL TRIAL: NCT06246825
Title: the Pathophysiology of the Onset of Atrial Fibrillation in Obstructive Sleep Apnea
Acronym: PARABOLA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Maarten van den Broek, Mr JLPM van den Broek, MD, Principal Investigator, Catharina Ziekenhuis Eindhoven
Other Study IDs: CatharinaZE_PARABOLA
Record Dates: First submitted 2023-12-07; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation; Obstructive Sleep Apnea of Adult
MeSH Terms: conditions — Atrial Fibrillation | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PARABOLA cohort: Patients with paroxysmal or persistent atrial fibrillation and a high likelihood of obstructive sleep apnea
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — Patients with a high likelihood of having obstructive sleep apnea will undergo a polysomnography, as recommended by the guidelines

SUMMARY:
Rationale: Obstructive sleep apnea (OSA) is a highly prevalent, often undiagnosed, modifiable risk factor for atrial fibrillation (AF), as well as AF-related complications and treatment effectiveness. It is unclear which OSA-related pathophysiological mechanism, i.e. intrathoracic pressure shifts, hypoxemia or sympathovagal imbalance, plays the most dominant role, and a better understanding of these mechanisms could provide valuable information in future diagnostic and therapeutic strategies in this population. Objective: The primary objective is to assess the role of OSA-related pathophysiological mechanisms in the initiation of AF by a multi-parametric strategy that combines the estimated parameters. The main hypothesis is that intrathoracic pressure fluctuations are the predominant mechanism. The secondary objective is to validate a nonobtrusive sensing technology based on photoplethysmography (PPG) and diaphragm electromyography (dEMG) measurements as surrogates for gold standard technology based on invasive intraoesophageal pressure (PES) measurement. Study population: Adult patients with paroxysmal AF with nocturnal onset and high risk of OSA based on the STOP-BANG questionnaire. Study design: An observational study in a selected cohort. Subjects are recruited from the AF outpatient clinic of the Catharina Hospital, and referred to Kempenhaeghe Centre for Sleep Medicine for a one-night full PSG, with the addition of dEMG and PPG. The acquired data will be analysed at the Eindhoven Technical University. Main study parameters/endpoints: Primary endpoint: Identification of prognostic factors for the initiation of AF in relation to OSA-related pathophysiological mechanisms..nl

ELIGIBILITY:
Inclusion Criteria:

Paroxysmal or persistent AF

AND

* STOP-BANG score >5 or STOP-BANG >4 and typical nocturnal onset of AF
* A positive WATCH-PAT screening
* very high clinical suspicion of OSA, with STOP-BANG score >3

Exclusion Criteria:

* current adequate treatment of OSA
* Reversible cause of AF
* severe lung disease (COPD Gold IV, pumonary fibrosis, lobectomy) wever esophageal disease (malignancy, stricture, esophagectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited in the Cardiology department of the Catharina Hospital Eindhoven (CZE). Patients presented here are referred by general practitioners and cardiologists in neighboring hospitals (Elkerliek Helmond, St. Anna Geldrop, St Jans Gasthuis Weert, Maxima Medisch Centrum Veldhoven, Bernhoven Uden). These patients generally have a high AF burden and frequent paroxysms. Patients with frequent paroxysms are preferred, as those have the highest chance of onset of AF during the one-night PSG. A large number of patients, approximately 400 unique patients per year, visits this clinic and, based on a small sample, 38% would meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory effort | 1 night, during the polysomnography
  Respiratory effort is measured by thoracoabdominal respiratory inductance plethysmography belts. We will calculate the integral/area above the curve of the amount of stretch on the belt (in mV) and the duration of inspiration (in seconds).
  Respiratory effort (mV*s) will be measured during baseline breathing (i.e. the awake period before sleep onset), during hazard periods (prior to onset of arrhythmia) and during control periods (same sleep stage as hazard period).
  Since respiratory effort is not standardized, the respiratory effort during control and hazard periods will be compared to baseline breathing (i.e. hazard period respiratory effort / baseline respiratory effort vs. control period / baseline respiratory effort)
Invasive respiratory effort | 1 night, during the polysomnography
  Invasive respiratory effort is measured by intraesophageal pressure sensor (Pes), if the patient tolerates this and can sleep with it. We will calculate the integral/area above the curve of the amount of pressure difference (in mmHg) and the duration of inspiration (in seconds).
  Respiratory effort (mmHg*s) will be measured during baseline breathing (i.e. the awake period before sleep onset), during hazard periods (prior to onset of arrhythmia) and during control periods (same sleep stage as hazard period).
  Since respiratory effort is not standardized, the respiratory effort during control and hazard periods will be compared to baseline breathing (i.e. hazard period respiratory effort / baseline respiratory effort vs. control period / baseline respiratory effort). Comparable to primary outcome 1
hypoxic burden | 1 night, during the polysomnography
  Blood oxygen levels (SpO2) are measured transcutaneously. Hypoxic burden will be calculated by calculating the integral of time (in seconds) and SpO2 < average SpO2, as published prior. The hypoxic burden beween hazard and control periods (see outcome 1 and 2) will be compared.
Vagal tone | 1 night, during the polysomnography
  The vagal tone will be assessed non-invasive through heart rate variability parameters (mainly LF/HF ratio (unitless) and RMSSD (ms^2). The heart rate variability parameters will be compared between hazard and control periods.

SECONDARY OUTCOMES:
Validation of diaphragm EMG | 1 night, during the polysomnography
  We will validate an algorithm that will try to assess the respiratory effort based of the signals of the diaphragm EMG by either using maximum amplitude (mV) or by combining the amplitude the signal (mV) with the duration (s)

CONTACTS AND LOCATIONS:
Overall Officials: Lukas RC Dekker, MD, PhD, prof, Study Chair — Eindhoven University of Technology / Catharina Hospital Eindhoven
Locations (1):
- Catharina Ziekenhuis, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonimized, full PSG data can be shared for scientific purposes only.
Supporting Information: Study Protocol, CSR
Time Frame: 20 years
Access Criteria: Purely scientific purposes only